CLINICAL TRIAL: NCT00711698
Title: PCA for Pain Control in Adults With Sickle Cell Disease in the Emergency Department (ED) Decreases Admission Rates Over Standard Bolus Therapy
Brief Title: Comparison of Patient Controlled Analgesia (PCA) Versus Bolus Narcotic Therapy for the Treatment of Vaso-Occlusive Crisis (VOC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: technical difficulties coordinating study
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00001163
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): In this arm patients will be randomized to receive a bolus of narcotic followed by PCA.
  Interventions: Procedure: Patient controlled analgesia
- 2 (Active Comparator): In this arm patients will be randomized to the current standard of care of bolus narcotic treatment.
  Interventions: Drug: nurse-administered intermittent IV bolus opioid therapy (NAIBOD)

INTERVENTIONS:
Procedure: Patient controlled analgesia — Patients in this arm will be treated with a bolus of narcotic followed by PCA
  Arms: 1
Drug: nurse-administered intermittent IV bolus opioid therapy (NAIBOD) — In this arm patients will receive the current standard of care of IV bolus narcotic therapy
  Arms: 2

SUMMARY:
This research is being done to find out the best way to give narcotics for pain relief in adults with sickle cell disease and painful crisis. This study is a comparison of two ways of giving narcotics. The first way is what occurs now in the Emergency Acute Care Unit (EACU) where patients are given a single intravenous (iv) dose of a narcotic which is repeated by the nurse as needed to control the pain. The second way is to provide a single iv dose of narcotic and then allow the patient to push a button and receive one or more additional doses of narcotic when he/she thinks it is needed. Our hypothesis is that PCA will be a more effective way of controlling pain.

ELIGIBILITY:
Inclusion Criteria:

* Documented sickle cell disease
* Signed consent in outpatient clinic or during a prior hospitalization
* 18+ years of age
* Seen in the ED with sickle cell pain crisis - this will be based on patients chief complaint that they are in a VOC.
* Requires IV administration of narcotics (has failed oral narcotic therapy at home)
* Must be 2 weeks since their last randomization on this study.

Exclusion Criteria:

* Contraindication to the use of IV narcotics
* Hypotension with systolic blood pressure (SBP) ≤ 90
* Respiratory rate ≤9
* Altered mental status
* Patient unable to understand how to use the PCA device
* Patient unwilling to use PCA device
* Pulse oximeter reading of ≤ 94% on room air
* Patient is allergic to IV morphine & hydromorphone & fentanyl.
* Patient is allergic to oral hydromorphone & morphine & oxycodone
* Patient has been randomized on this study 3 times before

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in admissions for those treated with a PCA in the ED v those that are given bolus narcotic dosing | Measured at time of discharge from ED

SECONDARY OUTCOMES:
Length of stay | Endpoints will be the time at which the decision for discharge from the EACU or transfer from the EACU to inpatient admission to the hospital is made
Total narcotic used | Endpoints will be the time at which the decision for discharge from the EACU or transfer from the EACU to inpatient admission to the hospital is made

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lanzkron, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States